CLINICAL TRIAL: NCT06941662
Title: HD Project: Neurodegenerative Disease Research Platform - Novel Remote Monitoring and Deep Phenotyping.
Brief Title: Huntington's Disease Biobank: Advancing Remote Monitoring and Deep Phenotyping
Status: Recruiting | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: Schwab Charitable Fund (Unknown)
Responsible Party: Principal Investigator, Kyan Younes, Assistant Professor, Stanford University
Other Study IDs: 74659
Record Dates: First submitted 2025-04-02; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Huntington Disease
Keywords: Huntington's disease biomarkers; remote monitoring; biobank; observational study
MeSH Terms: conditions — Huntington Disease | interventions — Blood Specimen Collection; Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, optional cerebrospinal fluid, optional skin biopsy, videos of motor exam, mobile app-based testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Huntington's disease: Individuals who carry the Huntington's disease mutation. Individuals with pre-manifest or manifest disease at all disease stages are welcome
  Interventions: Diagnostic Test: computer vision, remote monitoring, blood, urine, wrist bands, mobile-app

INTERVENTIONS:
Diagnostic Test: computer vision, remote monitoring, blood, urine, wrist bands, mobile-app — This is a low burden study that relies on a combination of cutting edge remote monitoring methods to deliver individualized evaluations to participants in their homes.

SUMMARY:
This observational study aims to identify novel biomarkers of disease onset and progression in Huntington's disease by integrating remote monitoring with fluid biomarkers. Using video-based computer vision and mobile app-based cognitive assessments combined with machine learning algorithms, we aim to develop markers that can be used by Huntington's disease patients at home.

Using machine learning to analyze videos of movement will capture the movements with an accuracy that will be as good as seeing an expert neurologist. These individualized markers can be followed over time to evaluate symptoms onset and change. The study will track disease progression and correlate these digital markers with changes in plasma and cerebrospinal fluid. The ultimate goal is to advance biomarker discovery and therapeutic development for Huntington's disease.

The study includes one in-person visit per year. A remote visit via Zoom or Facetime (15 min) every three months to record videos of movement. We can also share cutting-edge wristbands and a mobile phone app.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a positive test for the HD expansion mutation.

Exclusion Criteria:

* Individuals with movement disorders with a negative test for the HD expansion mutation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: community, neurology clinics, hospital, huntington's disease centers of excellence.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2035-12 (Estimated); Study Completion 2035-12 (Estimated)

PRIMARY OUTCOMES:
Unified Huntington's Disease Rating Scale (UHDRS) | Once a year in-person and 3 times a year remotely, until death or dropout of the study (average approximately 1 year)
  Neurological exam with a neurologist to document the motor exam

SECONDARY OUTCOMES:
Timed Up and Go (TUG) | Once a year in-person and 3 times a year remotely, until death or dropout of the study (average approximately 1 year)
  Timed stand from chair and walk
30-second Chair Stand Test | Once a year in-person and 3 times a year remotely, until death or dropout of the study (average approximately 1 year)
  Assesses lower body strength and endurance. Participants are instructed to stand up fully and sit back down as many times as possible within 30 seconds,

CONTACTS AND LOCATIONS:
Overall Officials: Kyan Younes, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No